CLINICAL TRIAL: NCT03649893
Title: The Effectivness of Multi-modal Intervention for Reducing Sedentary Behavior in Office Workers
Brief Title: Effectivness of Active Office Intervention
Acronym: ActiveOffice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Primorska (Other)
Collaborators: Innorenew CoE (Other)
Responsible Party: Principal Investigator, Nejc Sarabon, Assoc. Prof. Dr. Sc., University of Primorska
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Active Office
Record Dates: First submitted 2018-08-24; First posted 2018-08-28 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Sedentary Lifestyle
Keywords: sedentary behavior; phyical activity; workplace interventions; active breaks; workplace ergonomics
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will use conventional siiting-desk office.
- Active Office Group (Experimental): The experimental group will use active offfice, including sit-to-stand desk, bike desk, seddle chair and active breask.
  Interventions: Device: Active Office

INTERVENTIONS:
Device: Active Office — Active Office intervention includes sit-to-stand desk, bike desk, seddle chair, and active breaks.
  Arms: Active Office Group

SUMMARY:
The Active Office study is focusing on interventions with potential to reduce sedentary behavior and increase physical activity in office workers. The participants will be devided in two groups, the experimental and the control group. The participants in the experimental group will use active office (sit-to-stand desk, bike desk, seddle chair and active breaks) for one week, whereas the control group will remain in the conventional sitting-desk office. All the participants will wear ActivePal for 5 consecutive day and complete the measurements (heart rate, blood pressure). The goal of the study is to evaluate the effects of active office on sedentary behavior and physical activity levels in office workers.

DETAILED DESCRIPTION:
Sedentary behavior is racognised as an independent risk factor for the development of non-communicable diseases. It is estimated that office workers spent up to 80 % of their working time sedentary and do not compensate by sitting less in their leisure time. Therefore, interventions with potential to reduce sedentary behavior and increase phyical activity levels are of increasing interest. The aim of this study is to evaluate the effects of active office, including sit-to-stand desk, bike desk, seddle chair, and active breaks, on sedentary behavior, physical activity levels, and cardio-vascular parameters. The study design will be randomised control trial with one experimental and one control group. The participants in the experimental group will use active office for one week whereas the control group will use the conventional office. All the participants will wear ActivePal for 5 consecutive day and complete the measurements (heart rate, blood pressure). The participants will also complete quastionaires about the sedentary behavior and physical activity levels (Sedentary Behavior Questionnaire, Global Physical Activity Questionnaire). Moreover, at the baseline and on the last day of measurements the investigators will measure the work environment factors (light, noise, air flow, temperature). The goal of the study is to evaluate the effects of active office on sedentary behavior and physical activity levels in office workers.

ELIGIBILITY:
Inclusion Criteria:

* office workers spending at least 70 % of their working time sedentary
* aged between 18 and 65

Exclusion Criteria:

* body mass index > 30kg/m2
* pain presence in any musculokeletal part > 3 on 10-level scale
* presence of any non-communicable chronical diseases
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-05 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Weekly physical activity levels | 5 days
  Weekly physical activity levels will be measured with ActivePal sensors.
Weekly sitting time | 5 days
  Weekly sitting time will be measured with ActivePal sensors.

SECONDARY OUTCOMES:
Heart rate | 5 days
  Heart rate will be measured with Polar Heart Rate Monitor.
Blood Pressure | Baseline and after 5 days
  Blood pressure will be measured with electronic blood pressure monitor.
Global Physical Activity Questionnaire | Baseline and after 5 days
  Global Physical Activity Questionnaire is used to subjectively assess physical activity levels.
Sedentary Behavior Questionnaire | Baseline and after 5 days
  Sedentary Behavior Questionnaire is used to subjectively assess sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Sarabon, Phd, Principal Investigator — University of Primorska
Locations (1):
- InnoRenew, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: No